CLINICAL TRIAL: NCT03099824
Title: A Phase 1, Open-label Study to Compare the Safety and Pharmacokinetics of Various Formulations of Orally Administered Superoxide Dismutase Mimetic GC4711 With Intravenously Administered Superoxide Dismutase Mimetic GC4419 or GC4711 in Healthy Volunteers
Brief Title: A Phase 1 Study of the Safety and Pharmacokinetics of GC4711 (Oral Capsule) Compared to GC4419 (IV Infusion) and GC4711 (IV Infusion) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GTO-003
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — avasopasem manganese

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- GC4419 IV + GC4711 Oral G-101 (82mg) (Experimental)
  Interventions: Drug: GC4711 Oral Capsule G-101; Drug: IV GC4419
- GC4419 IV + GC4711 Oral G-101 (164mg) (Experimental)
  Interventions: Drug: IV GC4419; Drug: GC4711 Oral Capsule G-101
- GC4419 IV + GC4711 Oral G-101 (246mg) (Experimental)
  Interventions: Drug: IV GC4419; Drug: GC4711 Oral Capsule G-101
- GC4419 IV + GC4711 Oral G-111 (175mg) (Experimental)
  Interventions: Drug: IV GC4419; Drug: GC4711 Oral Capsule G-111
- GC4419 IV + GC4711 Oral G-112 (145mg) (Experimental)
  Interventions: Drug: IV GC4419; Drug: GC4711 Oral Capsule G-112
- GC4711 IV + GC4711 Oral G-119 (233mg) (Experimental)
  Interventions: Drug: GC4711 Oral Capsule G-119; Drug: IV GC4711
- GC4711 IV + GC4711 Oral G-125 (233mg) (Experimental)
  Interventions: Drug: GC4711 Oral Capsule G-125; Drug: IV GC4711

INTERVENTIONS:
Drug: GC4711 Oral Capsule G-101 — 82 mg (1 capsule)
  Arms: GC4419 IV + GC4711 Oral G-101 (82mg)
Drug: IV GC4419 — GC4419 will be infused IV as a single dose of 27 mg in 247 mL normal saline, totaling 250 mL, over a 60-minute period using a programmable pump.
  Arms: GC4419 IV + GC4711 Oral G-101 (164mg); GC4419 IV + GC4711 Oral G-101 (246mg); GC4419 IV + GC4711 Oral G-101 (82mg); GC4419 IV + GC4711 Oral G-111 (175mg); GC4419 IV + GC4711 Oral G-112 (145mg)
Drug: GC4711 Oral Capsule G-101 — 164 mg (2 capsules)
  Arms: GC4419 IV + GC4711 Oral G-101 (164mg)
Drug: GC4711 Oral Capsule G-101 — 246 mg (3 capsules)
  Arms: GC4419 IV + GC4711 Oral G-101 (246mg)
Drug: GC4711 Oral Capsule G-111 — 175 mg (1 capsule)
  Arms: GC4419 IV + GC4711 Oral G-111 (175mg)
Drug: GC4711 Oral Capsule G-112 — 145 mg (1 capsule)
  Arms: GC4419 IV + GC4711 Oral G-112 (145mg)
Drug: GC4711 Oral Capsule G-119 — 233 mg (1 capsule)
  Arms: GC4711 IV + GC4711 Oral G-119 (233mg)
Drug: GC4711 Oral Capsule G-125 — 233 mg (1 capsule)
  Arms: GC4711 IV + GC4711 Oral G-125 (233mg)
Drug: IV GC4711 — GC4711 will be infused IV as a single dose of 30 mg in 250 mL normal saline, totaling 251 mL, over a 60-minute period using a programmable pump.
  Arms: GC4711 IV + GC4711 Oral G-119 (233mg); GC4711 IV + GC4711 Oral G-125 (233mg)

SUMMARY:
The purpose of the phase 1, GTO-003 clinical study is to determine the safety and pharmacokinetics of a single dose of a new drug called GC4711 when given as an oral capsule. This study will compare capsules of GC4711 when given orally to a similar drug, GC4419, or GC4711 when either is given as an intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between 18 and 50 years (inclusive) of age;
2. Subjects who provide written informed consent
3. Body Mass Index (BMI) 18 to 32 kg/m2 (inclusive) and weighing at least 50 kg during Screening and at Baseline. Every effort will be made to enroll across BMI range to evaluate relation between dose and weight;
4. Subjects in general good health in the investigator's opinion
5. Chest X-ray free of clinically significant abnormalities
6. Blood pressure and heart rate within normal limits
7. Female subjects must:

   1. Have a negative serum pregnancy test during Screening and a negative urine pregnancy test at Baseline, and be willing and able to use a medically acceptable method of birth control or be postmenopausal.
   2. Be non-lactating
   3. Be at least two years postmenopausal, surgically sterile or practicing effective contraception

Exclusion Criteria:

1. History of clinically significant illness, medical condition, or laboratory abnormality within three months
2. History of any clinically significant cardiovascular, hepatic, renal, or gastrointestinal abnormality;
3. History of hypotension
4. Known contraindication, hypersensitivity and/or allergy to investigational products
5. Use of any prescription or over-the-counter medication within one week prior to baseline;
6. Anticipated need for any medication during the course of the study
7. Use of nitrates or erectile dysfunction drugs such as phosphodiesterase type 5 (PDE 5) inhibitors (e.g., sildenafil, tadalafil, or similar agents), from 24 hours prior to screening throughout participation in the study;
8. Use of or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure
9. Presence of orthostatic hypotension at screening or baseline
10. Use of any vitamin or mineral supplement 24 hours prior to dosing, or anticipated use of any vitamin or mineral supplement throughout the duration of the study;
11. Positive HIV, Hepatitis B or Hepatitis C serology at Screening;
12. Known history of substance abuse, drug addiction, or alcoholism within 3 years
13. Anticipated inability to abstain from alcohol, tobacco, or caffeine use from 48 hours prior to the administration of study drug and throughout the duration of the study;
14. Positive drug and alcohol toxicology screens during Screening and at Baseline;
15. History of smoking or any use of a tobacco product within six months prior to Baseline;
16. Donation of blood or blood products within 30 days prior to the Baseline and through duration of study;
17. Mentally unstable or incapable of being compliant with the protocol
18. Receipt of an investigational test substance within three months prior to the first dose of investigational products (GC4419, GC4711, or placebo), or anticipated receiving any investigational products (including placebo on another investigational study) other than GC4711 and GC4419 during the course of this study;
19. Subject has previously participated in this study, or in a prior study of GC4419, GC4711 or GC4702.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Laboratory Abnormalities | From randomization through study completion (estimated up to 13 days)
  Number of Participants With Treatment-Emergent Adverse Events and/or Laboratory Abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Chief Medical Officer
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No